CLINICAL TRIAL: NCT00395226
Title: "Zinc Sulfate in the Treatment of Rosacea: A Randomized, Controlled Trial." Prospective, Double Blind, Randomized, Controlled Trial Comparing the Effects of Supplemental Zinc Sulfate and Placebo on the Severity of Rosacea.
Brief Title: Zinc Sulfate in the Treatment of Rosacea: A Randomized, Controlled Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting subjects
Sponsor: Essentia Health (Other)
Responsible Party: Joel Bamford, MD, St. Mary's duluth Clinic Health System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-05-03
Record Dates: First submitted 2006-10-31; First posted 2006-11-02 (Estimated); Results first posted 2011-06-30 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Rosacea
Keywords: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zinc sulfate (Experimental): 220 mg of zinc sulfate
  Interventions: Drug: zinc sulfate
- Lactose (Placebo Comparator): 270 mg lactose
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: zinc sulfate — zinc sulfate 220 mg bis for 90 days
  Arms: Zinc sulfate
Drug: placebo — placebo bid for 90 days
  Arms: Lactose

SUMMARY:
Rosacea is a common chronic dermatological condition, characterized by recurrent or persistent redness, permanent dilation of small blood vessel causing small red lesions, and papules/pustules. The signs of rosacea are usually confined to the face, but may appear on the neck, scalp or trunk. Opthalmologic findings are also common. Rosacea is usually described as being most common in fair skinned women over 40. The purpose of the study is to determine whether oral Zinc Sulfate treatment is an effective treatment for facial rosacea.

DETAILED DESCRIPTION:
Rosacea is a common chronic dermatological condition. The epidemiology of rosacea has not been determined extensively, due to part in problems with case definition. Rosacea is usually described as being most common in fair skinned women over the age of 40. However it occurs in most adult populations, including both men and women of all ages, and in people of many complexion types, including African Americans and Asians.

Although rosacea is encountered frequently in primary care and dermatology practices, its precise incidence and prevalence are not known. The etiology and pathogenesis of rosacea are unknown. Both genetic and environmental factors are thought to be important. A wide range of medical and surgical interventions have been used in the management of rosacea, including dietary management, topical and systemic antibiotics, azelaic acid, low dose isotretinoin, and laser treatments for telangiectasia and rhinophyma. No single regimen has been found to be entirely satisfactory.

Zinc has been found to be effective in managing several dermatological conditions, especially acne. It has also been found to be of benefit in dermatological conditions such as viral warts and cutaneous leishmaniasis.

No studies have been published on the use of Zinc in the treatment of rosacea. This will be a prospective, double blind, randomized, controlled trial, comparing the effects of supplemental and placebo on the severity of rosacea. Enrolled subjects will be assigned to one of two study arms.

Subjects and investigators will be blinded regarding treatment. After evaluation, meeting the study criteria,obtaining informed consent, and initiating study related procedures, the subject will take oral study drug or placebo, bid, for 90 days.

Subjects are followed via phone call at one week and 6 weeks after enrollment into the study. At the conclusion of the 90 day study, subjects will be re-examined.

The primary endpoint of this study will be the severity of rosacea at the end of the 90 day intervention period.

The efficacy of Zinc vs. placebo will be assessed by a comparison of the change in the severity of rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of facial rosacea made or confirmed by one of the investigators.
* Severity of signs of rosacea "greater than mild" at the time of enrollment.

Exclusion Criteria:

* Treatment for rosacea during the 3 months prior to enrollment.
* Use of zinc dietary supplement > 25 mg per day during the 3 months prior to enrollment ( Most patients taking multivitamins with Zinc, often 15 mg per day, will not be excluded, whereas most patients taking additional Zinc supplements, often 25-50 mg per day or more will be excluded.)
* Diagnosis of rosacea fulminancy.
* Pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2006-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Bamford, MD, Principal Investigator — Essentia Health
Locations (1):
- St. Mary's Duluth Clinic Health System, Duluth, Minnesota, United States

REFERENCES:
- [Background] Berg M, Liden S. An epidemiological study of rosacea. Acta Derm Venereol. 1989;69(5):419-23. PMID 2572109
- [Background] Bamford JT. Rosacea: current thoughts on origin. Semin Cutan Med Surg. 2001 Sep;20(3):199-206. doi: 10.1053/sder.2001.27553. PMID 11594675
- [Background] Millikan L. The proposed inflammatory pathophysiology of rosacea: implications for treatment. Skinmed. 2003 Jan-Feb;2(1):43-7. doi: 10.1111/j.1540-9740.2003.01876.x. PMID 14673323
- [Background] Wilkin JK. Rosacea. Pathophysiology and treatment. Arch Dermatol. 1994 Mar;130(3):359-62. doi: 10.1001/archderm.130.3.359. No abstract available. PMID 8129416
- [Background] Thiboutot DM. Acne and rosacea. New and emerging therapies. Dermatol Clin. 2000 Jan;18(1):63-71, viii. doi: 10.1016/s0733-8635(05)70147-9. PMID 10626112
- [Background] Bikowski JB.Del Rosso JQ, Goldberg DJ, Margolis DJ, Van Zuuren EJ, Wolf JE. Future Trends in the Treatment of Rosacea. Cutis. 2005;75(Suppl 3):33-36
- [Background] Tuleya S. Research Highlights: Acne and Rosacea Treatments. Skin and Agining.2003;11(8):70-72.
- [Background] Fraker PJ, King LE. Reprogramming of the immune system during zinc deficiency. Annu Rev Nutr. 2004;24:277-98. doi: 10.1146/annurev.nutr.24.012003.132454. PMID 15189122
- [Background] Fraker PJ, King LE, Laakko T, Vollmer TL. The dynamic link between the integrity of the immune system and zinc status. J Nutr. 2000 May;130(5S Suppl):1399S-406S. doi: 10.1093/jn/130.5.1399S. PMID 10801951
- [Background] Walker CF, Black RE. Zinc and the Risk for Infectious Disease. ann Intern Med. 1996;125(2):81-88.
- [Background] Mossad SB, Macknin ML, Medendorp SV, Mason P. Zinc gluconate lozenges for treating the common cold. A randomized, double-blind, placebo-controlled study. Ann Intern Med. 1996 Jul 15;125(2):81-8. doi: 10.7326/0003-4819-125-2-199607150-00001. PMID 8678384
- [Background] ___.What's New about Zinc. UC Berkeley Wellness Letter. 2004:130:1344S-1349S.
- [Background] Hambidge M. Human zinc deficiency. J Nutr. 2000 May;130(5S Suppl):1344S-9S. doi: 10.1093/jn/130.5.1344S. PMID 10801941
- [Background] Hoffman HN 2nd, Phyliky RL, Fleming CR. Zinc-induced copper deficiency. Gastroenterology. 1988 Feb;94(2):508-12. doi: 10.1016/0016-5085(88)90445-3. PMID 3335323
- [Background] Salzman MB, Smith EM, Koo C. Excessive oral zinc supplementation. J Pediatr Hematol Oncol. 2002 Oct;24(7):582-4. doi: 10.1097/00043426-200210000-00020. PMID 12368702
- [Background] Irving JA, Mattman A, Lockitch G, Farrell K, Wadsworth LD. Element of caution: a case of reversible cytopenias associated with excessive zinc supplementation. CMAJ. 2003 Jul 22;169(2):129-31. PMID 12874162
- [Background] Chandra RK. Excessive intake of zinc impairs immune responses. JAMA. 1984 Sep 21;252(11):1443-6. PMID 6471270
- [Background] Barceloux DG. Zinc. J Toxicol Clin Toxicol. 1999;37(2):279-92. doi: 10.1081/clt-100102426. PMID 10382562
- [Background] Schosinsky KH, Lehmann HP, Beeler MF. Measurement of ceruloplasmin from its oxidase activity in serum by use of o-dianisidine dihydrochloride. Clin Chem. 1974 Dec;20(12):1556-63. No abstract available. PMID 4214636
- [Background] West EC, Prohaska JR. Cu,Zn-superoxide dismutase is lower and copper chaperone CCS is higher in erythrocytes of copper-deficient rats and mice. Exp Biol Med (Maywood). 2004 Sep;229(8):756-64. doi: 10.1177/153537020422900807. PMID 15337829
- [Background] Dreno B, Amblard P, Agache P, Sirot S, Litoux P. Low doses of zinc gluconate for inflammatory acne. Acta Derm Venereol. 1989;69(6):541-3. PMID 2575335
- [Background] Dreno B, Moyse D, Alirezai M, Amblard P, Auffret N, Beylot C, Bodokh I, Chivot M, Daniel F, Humbert P, Meynadier J, Poli F; Acne Research and Study Group. Multicenter randomized comparative double-blind controlled clinical trial of the safety and efficacy of zinc gluconate versus minocycline hydrochloride in the treatment of inflammatory acne vulgaris. Dermatology. 2001;203(2):135-40. doi: 10.1159/000051728. PMID 11586012
- [Background] Chu A, Huber FJ, Plott RT. The comparative efficacy of benzoyl peroxide 5%/erythromycin 3% gel and erythromycin 4%/zinc 1.2% solution in the treatment of acne vulgaris. Br J Dermatol. 1997 Feb;136(2):235-8. PMID 9068739
- [Background] Meynadier J. Efficacy and safety study of two zinc gluconate regimens in the treatment of inflammatory acne. Eur J Dermatol. 2000 Jun;10(4):269-73. PMID 10846252
- [Background] Schachner L, Eaglstein W, Kittles C, Mertz P. Topical erythromycin and zinc therapy for acne. J Am Acad Dermatol. 1990 Feb;22(2 Pt 1):253-60. doi: 10.1016/0190-9622(90)70034-f. PMID 2138176
- [Background] Verma KC, Saini AS, Dhamija SK. Oral zinc sulphate therapy in acne vulgaris: a double-blind trial. Acta Derm Venereol. 1980;60(4):337-40. doi: 10.2340/0001555560337340. PMID 6163281
- [Background] Al-Gurairi FT, Al-Waiz M, Sharquie KE. Oral zinc sulphate in the treatment of recalcitrant viral warts: randomized placebo-controlled clinical trial. Br J Dermatol. 2002 Mar;146(3):423-31. doi: 10.1046/j.1365-2133.2002.04617.x. PMID 11952542
- [Background] Sharquie KE, Najim RA, Farjou IB, Al-Timimi DJ. Oral zinc sulphate in the treatment of acute cutaneous leishmaniasis. Clin Exp Dermatol. 2001 Jan;26(1):21-6. doi: 10.1046/j.1365-2230.2001.00752.x. PMID 11260171
- [Background] Berne B, Venge P, Ohman S. Perifolliculitis capitis abscedens et suffodiens (Hoffman). Complete healing associated with oral zinc therapy. Arch Dermatol. 1985 Aug;121(8):1028-30. PMID 4026339
- [Background] Rostan EF, DeBuys HV, Madey DL, Pinnell SR. Evidence supporting zinc as an important antioxidant for skin. Int J Dermatol. 2002 Sep;41(9):606-11. doi: 10.1046/j.1365-4362.2002.01567.x. PMID 12358835
- [Background] Dreno B, Trossaert M, Boiteau HL, Litoux P. Zinc salts effects on granulocyte zinc concentration and chemotaxis in acne patients. Acta Derm Venereol. 1992 Aug;72(4):250-2. PMID 1357876
- [Background] Wilkin J, Dahl M, Detmar M, Drake L, Liang MH, Odom R, Powell F; National Rosacea Society Expert Committee. Standard grading system for rosacea: report of the National Rosacea Society Expert Committee on the classification and staging of rosacea. J Am Acad Dermatol. 2004 Jun;50(6):907-12. doi: 10.1016/j.jaad.2004.01.048. No abstract available. PMID 15153893

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 65 participants were recruited between August 2006 and April 2008
Pre-assignment Details: 65 participants were assessed for eligibility. 12 did not meet inclusion criteria (severity of facial rosacea "greater than mild" at the time of enrollment, at least 5 of 12 on the Modified Rosacea Severity Scoring System).
Period: Overall Study
Arm/Group | Placebo (Lactose) | Zinc Sulfate
Started | 26 | 27
Completed | 22 | 22
Not Completed | 4 | 5
Not completed — Adverse Event | 4 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Lactose) | Zinc Sulfate | Total
Number analyzed (Participants) | 26 | 27 | 53
Age Continuous [Mean (Standard Deviation); unit: years] | 47.3 (13.4) | 52.8 (10.5) | 50.1 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 7 | 7 | 14
Race/Ethnicity, Customized [Number; unit: participant]
  Caucasian | 24 | 26 | 50
  Non-Caucasian | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 26 | 27 | 53
Length of Rosacea [Number; unit: participant]
  < 1 year | 1 | 2 | 3
  1-2 years | 0 | 3 | 3
  2-5 years | 12 | 4 | 16
  5-10 years | 4 | 10 | 14
  > 10 years | 9 | 8 | 17
Rosacea Severity Score [Mean (Standard Deviation); unit: units on scale 0 to 12] — Modified Rosacea Severity Scoring System evaluating four signs of rosacea, flushing (transient erythema or redness), erythema (redness), papules and pustules and telangiectasia (spider-veins) ranges from 0 (best, absent) to 12 (worst, severe on all items)
  units on scale 0 to 12 | 6.8 (1.4) | 6.3 (1.2) | 6.5 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Severity of Facial Rosacea After 90 Days of Treatment
Description: Modified Rosacea Severity Scoring System evaluating four signs of rosacea, flushing (transient erythema or redness), erythema (redness), papules and pustules and telangiectasia (spider-veins) ranges from 0 (best, absent) to 12 (worst, severe on all items)
Time Frame: 90 days
Measure: Mean (95% Confidence Interval); unit: units on scale 0 to 12
Arm/Group | Placebo (Lactose) | Zinc Sulfate
Number analyzed (Participants) | 22 | 22
units on scale 0 to 12 | 4.9 [4.1 to 5.6] | 5.1 [4.2 to 6.0]
Statistical Analysis 1: Comparison: Placebo (Lactose) vs Zinc Sulfate; The null hypothesis was "no group differences." The alternative hypothesis was that the zinc sulfate arm is superior to placebo arm; Test type: Superiority or Other; p = 0.2840, ANCOVA — The a priori significance threshold level was 0.05 (two-sided); The ANCOVA used group as a factor and baseline rosacea severity score as a covariate; Mean Difference (Final Values) = 0.57, 95% CI 2-sided [-0.47 to 1.62] — The effect of zinc sulfate treatment on rosacea severity score was estimated with baseline rosacea severity score included in the regression model

ADVERSE EVENTS:
Arm/Group | Placebo (Lactose) | Zinc Sulfate
Serious Adverse Events (participants affected / at risk) | 0 | 2
Other Adverse Events (participants affected / at risk) | 15/25 | 15/27
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Placebo (Lactose) | Zinc Sulfate
Allergic reaction (Skin and subcutaneous tissue disorders) | 0/25 (0) | 1/27 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0/25 (0) | 1/27 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Lactose) (N=25) | Zinc Sulfate (N=27)
gastrointestinal disorders (Gastrointestinal disorders) | 12 | 15 — stomach upset, including nausea, discomfort, gas, diarrhea, constipation, and increased bowel movements
rosacea outbreak (Skin and subcutaneous tissue disorders) | 3 | 0 — including redness and itching

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes